CLINICAL TRIAL: NCT05755958
Title: Doubled Blind Evaluation of the Efficacy of High Intensity Focused Ultrasound (HIFU) Treatment on Symptoms in Patients Treated for Rectal Endometriosis Compared to Sham.
Brief Title: Evaluation of the Efficacy of HIFU Treatment on Rectal Endometriosis Symptoms.
Acronym: ENDO-HIFU-R2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIFU/F/21.12
Record Dates: First submitted 2023-01-30; First posted 2023-03-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
Keywords: Rectal Endometriosis; HIFU; FocalOne; High Intensity Focused Ultrasound
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIFU SHAM (Sham Comparator): The patient placed in the right lateral decubitus position under general anesthesia or spinal anesthesia on the operating table. An endorectal probe is inserted in the patient's rectum. The probe includes an imaging transducer to visualize the endometriosis lesions and locate areas to be treated and an ultrasound therapy transducer to administer the HIFU treatment. After identification of the treatment area, HIFU shots will not be delivered on the lesion to be treated in a blinded manner.
  Patients randomized to this arm will received exactly the same procedure as patients in the HIFU group with the exception of the HIFU shots.
  Interventions: Device: SHAM HIFU procedure
- HIFU TREATMENT (Active Comparator): The patient placed in the right lateral decubitus position under general anesthesia or spinal anesthesia on the operating table. An endorectal probe is inserted in the patient's rectum. The probe includes an imaging transducer to visualize the endometriosis lesions and locate areas to be treated and an ultrasound therapy transducer to administer the HIFU treatment. After identification of the treatment area, HIFU shots will be delivered on the lesion to be treated in a blinded maner.
  Interventions: Device: HIFU treatment in rectal Endometriosis

INTERVENTIONS:
Device: HIFU treatment in rectal Endometriosis — HIFU treatment of rectal endometriosis
  Arms: HIFU TREATMENT
Device: SHAM HIFU procedure — SHAM HIFU procedure
  Arms: HIFU SHAM

SUMMARY:
Rectal endometriosis (RE) induces lesions associated with painful symptoms that can alter quality of life. High Intensity Focused Ultrasound (HIFU) is a non-invasive ablative procedure using a high-intensity ultrasound probe to induce tissue devitalization using acoustic cavitation and thermal ablation.

Focal One® is a transrectal HIFU device, which is validated to treat prostatic cancer.

In this comparative, randomized, double blind study , the primary objective is to evaluate the efficacy of the HIFU treatment of rectal endometriosis with Focal One® HIFU device on the Acute Pelvic Pain 3 months after HIFU treatment, in comparison to a Sham group.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older,
* Rectal endometriosis on preoperative imaging with no other digestive location,
* Symptomatic patient (Acute pelvic pain > 3), in failure of drug treatment,
* Endometriotic lesion visible on ultrasound and confirmed on MRI,
* Centralized MRI, reviewed and validated by the MRI review committee,
* No current pregnancy and no pregnancy plan during the study period,
* Patient agreeing not to change her hormonal treatment throughout the study period,
* Patient accepting the constraints of follow-up defined in the framework of the study,
* Patient affiliated to French health insurance.

Exclusion Criteria:

* Ongoing urogenital infection,
* Anorectal anatomy incompatible with HIFU treatment,
* Overall pain level considered intolerable by the patient and making a potential 3-months delay management impossible,
* History of segmental rectal resection or discoid resection,
* Patient with an implant located less than 1 cm from the treatment area,
* Inflammatory disease of the colon,
* Allergy to latex,
* No scheduled endometriosis procedures during study follow-up,
* Treatment of endometriosis in the context of pregnancy desire for which a 3-month delay is not appropriate
* Patient with contraindications to MRI,
* Patient who has already received HIFU treatment for a rectal endometriotic lesion,
* Patient who does not speak or read French,
* Patient deprived of liberty following a judicial or administrative decision,
* Patient in labor or nursing,
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the evolution in the level of acute pelvic pain compared to the sham intervention group. | 3 months
  The efficacy of HIFU treatment will be assessed by comparing the evolution in the level of acute pelvic pain assessed by Visual Analog Scale (VAS), ranging from 0 (best situation) to 10 (worst situation) at 3 months, to the pre-treatment pain level. The evolution in the HIFU group will be compared to those in the sham intervention group.

SECONDARY OUTCOMES:
Adverse Events occurrence and comparison between the two groups | 3 months
  Occurrence of adverse events during the 3 months of post-intervention follow-up will be evaluated in each group.
Symptoms evolution evaluation | 1 and 3 months
  The Visual Analog Scale (VAS) symptoms questionnaire to assess gynecologic, digestive, urinary and general symptoms though 15 different visual scales ranging from 0 (representing no symptom) to 10 (representing the worst patient feeling).
  Symptoms level will be collected before treatment and at 1 and 3 months after treatment. The symptoms' evolution in the HIFU group will be compared to those in the sham intervention group.
Evaluation of anal continence | 1 and 3 months
  The Wexner total score ranges from 0 to 23 points corresponding to the sum of the 6 questions. Anal incontinence is considered as mild for a total score from 0 to 4, moderate when ranging from 5 to 9, important from 10 to 16, and considered as severe if equal to 16 or higher.
  Symptoms level will be collected before treatment and at 1 and 3 months after treatment. The symptoms' evolution in the HIFU group will be compared to those in the sham intervention group.
Evaluation of constipation | 1 and 3 months
  The KESS (Knowles-Eccersley-Scott Symptom) question is composed of the sum of 11 questions evaluating constipation. The total score ranges from 0 to 39 points corresponding to a total constipation status. Constipation is generally defined as a score above 10.
  Symptoms level will be collected before treatment and at 1 and 3 months after treatment. The symptoms' evolution in the HIFU group will be compared to those in the sham intervention group.
Evaluation of urinary symptoms | 1 and 3 months
  USP (Urinary Symptoms Profile) is a questionnaire that assesses urinary symptoms. It includes 13 questions grouped in 3 domains:
  * Incontinence ranging from 0 to 9
  * Overactive bladder ranging from 0 to 21
  * Dysuria ranging from 0 to 9
  The USP total score is the sum of all the 13 answers and ranges from 0 to 39 points, where 39 corresponds to the worst situation. Urinary dysfunction is generally defined as a score above 10.
  Symptoms level will be collected before treatment and at 1 and 3 months after treatment. The symptoms' evolution in the HIFU group will be compared to those in the sham intervention group.
Evaluation of sexual fonction | 1 and 3 months
  FSFI (Female Sexual Function Index scoring) is a validated questionnaire, including 19 items, which assesses different domains of sexual function (desire, arousal, lubrication, orgasm, satisfaction, and pain) in addition to providing an overall score regarding sexual function. FSFI total score ranges from 2 (worst situation) to 36 (best situation).
  Symptoms level will be collected before treatment and at 1 and 3 months after treatment. The symptoms' evolution in the HIFU group will be compared to those in the sham intervention group.
Quality of life evoluation | 1 and 3 months
  The questionnaire for the Quality of life evaluation is MOS-SF-36 (Medical Outcomes Study Short Form 36 item Health survey).
  The MOS-SF-36 questionnaire consists of 36 questions which are divided into 8 different domains. Each domain is represented by the average of several questions (after recoding). Two scores, physical and mental, are then calculated. The maximum value of 100 corresponds to an optimal quality of life as described by the patient and zero the worst situation.
  Quality of life will be collected before treatment and at 1 and 3 months after treatment. The quality of life evolution in the HIFU group will be compared to those in the sham intervention group.
Volume lesion evaluation | 3 months
  The volume of endometriosis nodule will be evaluated on MRI, before treatment and at 3 months after treatment.
  (blinded evaluation of the treatment groups). The volume variation observed in the HIFU group will be compared with those observed in the Sham Intervention group.
Post treatment medication rate | 10 days
  The level of post-treatment medication during the first 10 days will be collected in the patient diary. The level of post-treatment medication in HIFU group will be compared to those in the sham intervention group.
Post treatment pain rate | 10 days
  The level of pain will be evaluated by daily self-evaluation by the patients;rom 0 (best situation) to 10 (worst situation), and collected on the daily diary during the first 10 days post-intervention. The pain level in HIFU group will be compared to the sham intervention group.
Overall recovery time evaluation | 3 months
  The overall recovery time will be evaluated by the patients on the patient diary.
  The overall recovery time observed in the HIFU group will be compared to those observed in the Sham intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Dubernard, Pr, Principal Investigator — EDAP TMS
Locations (9):
- France (9):
  - Hopital Privé de Provence, Aix-en-Provence
  - CHU de Angers, Angers
  - Clinique Tivoli-Ducos, Bordeaux
  - Chu Estaing, Clermont-Ferrand
  - Hôpital du Kremlin Bicetre, Le Kremlin-Bicêtre
  - Hôpital privé Le Bois, Lille
  - Hopital de la Croix Rousse, Lyon
  - Hôpital COCHIN, Paris
  - CHU Strasbourg, Strasbourg